CLINICAL TRIAL: NCT02610855
Title: Effect of Treatment on Activity and Muscle Function in Pediatric Patients With Scoliosis (SAMUS SCOLI)
Brief Title: Effect of Treatment on Activity and Muscle Function in Pediatric Patients With Scoliosis
Acronym: SAMUS SCOLI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Todd A. Milbrandt, M.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-005602
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Spinal Fusion Surgery (Active Comparator): The surgical participants recruited from the pediatric orthopaedic clinic and have severe scoliosis curves requiring posterior spinal fusion. Physical activity measured using Tri-axial accelerometers and paraspinal muscle stiffness measured by Shear Wave Elastography (SWUE) ultrasound will be quantified before and one year after spinal fusion surgery.
  Interventions: Procedure: Spinal Fusion Surgery; Device: Tri-axial Accelerometers; Other: Shear Wave Elastography (SWUE)
- Brace Treatment (Active Comparator): The bracing participants have scoliosis curves that require treatment with a spinal brace for at least the next year. All braces will have monitors to record hours of brace wear, as is current standard of care. Physical activity measured using Tri-axial accelerometers and paraspinal muscle stiffness measured by Shear Wave Elastography (SWUE) ultrasound will be quantified before bracing and after one year.
  Interventions: Other: Bracing; Device: Tri-axial Accelerometers; Other: Shear Wave Elastography (SWUE)
- Control Arm (Other): The control group are participants who do not have scoliosis. Physical activity measured using Tri-axial accelerometers and paraspinal muscle stiffness measured by Shear Wave Elastography (SWUE) ultrasound will be quantified at baseline and one year after enrollment.
  Interventions: Device: Tri-axial Accelerometers; Other: Shear Wave Elastography (SWUE)

INTERVENTIONS:
Procedure: Spinal Fusion Surgery — Participants with severe scoliosis curves requiring spinal fusion surgery.
  Arms: Spinal Fusion Surgery
Other: Bracing — Participants with scoliosis curves that require brace treatment for at least the next year. Braces include monitors to record hours of brace wear, as is current standard of care.
  Arms: Brace Treatment
Device: Tri-axial Accelerometers — Four monitors are place on the participant (waist, thigh, both ankles), attached with straps. Periods of static and dynamic activity are measured based on accelerations in three orthogonal directions for 4 day's time while participating in regular daily activities.
  Other Names: ActiGraph GT3X+
Other: Shear Wave Elastography (SWUE) — SWUE is an ultrasound technique for noninvasively evaluating the mechanical properties (stiffness) of skeletal muscle tissue. A commercial ultrasound scanner (Aixplorer from Supersonic Imagine, France) with 2D real time SWUE will be used. The Aixplorer uses ultrasonic push beams to produce shear waves in tissue. The shear wave propagation speed is inherently related to tissue mechanical properties and is used to create a quantitative 2D elastogram of the tissue.

SUMMARY:
This study will explore the relationship between skeletal muscle and physical activity in scoliosis patients to provide insight into both the etiology of scoliosis and potential ways to mitigate the potential harms of treatment.

DETAILED DESCRIPTION:
The aims include first, to quantify the posture and physical activity of patients in the community before and after scoliosis treatment and compare to age-matched controls. Patients undergoing bracing or surgery for scoliosis will wear novel low-profile electronic monitors for 4 days prior to and at one year after initiation of treatment. Accelerometer data from the 4 activity monitors are combined for a comprehensive profile of daily activity, above and beyond that of a typical pedometer. Analysis will show a participant's % active time vs. static, % time sitting vs. lying down vs. standing vs. walking, total number of steps taken per day, and cadence of walking during each activity bout. The amount of total daily time spent lying, sitting, standing, walking and running will be quantified using specialized processing algorithms developed at Mayo Clinic. Results will be compared to a group of age- and BMI-matched control patients with healed forearm fractures.

Second, to determine changes in the mechanical properties of the paraspinal skeletal musculature (muscles along the spine) in scoliosis patient before and after treatment with brace or spinal surgery.

Shear Wave Elastography (SWUE) is a technique that uses ultrasound, a non-invasive imaging technique, to detect mechanical properties of tissues. Using SWUE, the stiffness in the paraspinal muscles will be obtained by acquiring Shear modulus measurements, reported in kilo Pascal (kPa) units. 10 measurements will be obtained for each muscle and a region of interest (ROI) will be placed in the displayed elastogram or color map from each measurement to obtain a "kPa" value. A mean shear modulus or stiffness will be obtained by averaging all 10 results. The measurements from each ROI are derived using software built in the ultrasound equipment.

The change in paraspinal skeletal muscle stiffness will be assessed and compared to normal controls to determine characteristics of spinal musculature in scoliosis patients and the impact of treatment with bracing or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 9 to16 years of age
* Scoliosis/Surgery group; has severe scoliosis curves requiring posterior spinal fusion surgery
* Scoliosis/Brace group; has scoliosis curves requiring brace treatment for at least the next year
* The Control group will be aged matched participants who have healed forearm fractures and will be matched to case patients by age, gender, and Body Mass Index (BMI). These children will be considered normal subjects for both the accelerometers and the Shear Wave Elastography (SWUE)

Exclusion Criteria:

- Patients with underlying muscle conditions or neuromuscular scoliosis

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of day with static activity | Baseline, 1 year
  Physical activity is measured by 4 wearable Tri-axial Accelerometers, worn for a 4 day period at baseline (prior to surgery or brace placement) and at one year after surgery of brace placement. Each second of data will be classified as static or dynamic. Among static postures, lying, standing and sitting are determined based on the orientation of the waist and thigh accelerometers in relation to the line of gravity. Accelerometer data from the 4 activity monitors are combined to provide a total percentage of time with static activities.
Change in dynamic physical activity as measured by step counts | Baseline, 1 year
  Physical activity is measured by 4 wearable Tri-axial Accelerometers worn for a 4 day period at baseline (prior to surgery or brace placement) and at one year after surgery of brace placement. Each second of data will be classified as static or dynamic. Dynamic movements will be classified as walking, jogging or stair climbing based activity that exceeds the pre-defined accelerometer amplitude threshold. Step counts will be calculated based on detection of peak accelerations of the bilateral ankles using adaptive thresholds during the longest period of walking. Accelerometer data from the 4 activity monitors are combined to provide a total measure of dynamic physical activity.

SECONDARY OUTCOMES:
Change in mean paraspinal muscle stiffness | Baseline, 1 year
  Muscle stiffness is measured by Shear Wave Elastography (SWUE). This measurement evaluates normal muscle's passive and active properties at a variety of angles and tensions, resulting in a shear modulus reading, measured in average kilo Pascal units from 10 images of each muscle region of interest. A transducer is used with ultrasound to produce shear waves in tissue. The wave speed relates to the tissue's mechanical properties and is used to create a quantitative 2D elastogram of the tissue. Multiple shear modulus measurements will be averaged, and obtained:
  * on control subjects at the left and right sides of the T12 spine segment level
  * on the scoliosis patients, at the periapical area (apex of curve, where it is most tilted)
  * at the concave and convex sides as well as at an area remote from the curvature

CONTACTS AND LOCATIONS:
Overall Officials: Todd Milbrandt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials